CLINICAL TRIAL: NCT01161602
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Pharmacodynamics of Multiple Dose Levels of Pumosetrag in Patients With Symptoms Associated With Gastroesophageal Reflux Disease (GERD) Receiving a Standard Refluxogenic Meal
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacodynamics of Pumosetrag in Patients With Gastroesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edusa Pharmaceuticals, Inc. (Industry)
Other Study IDs: Pumo-10-001
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Symptoms of Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pumosetrag

ARMS (4):
- 0.2mg Pumosetrag (Experimental)
  Interventions: Drug: Pumosetrag
- 0.5mg Pumosetrag (Experimental)
  Interventions: Drug: Pumosetrag
- 0.8mg Pumosetrag (Experimental)
  Interventions: Drug: Pumosetrag
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pumosetrag
  Arms: 0.2mg Pumosetrag
Drug: Pumosetrag
  Arms: 0.5mg Pumosetrag
Other: Placebo
  Arms: Placebo
Drug: Pumosetrag
  Arms: 0.8mg Pumosetrag

SUMMARY:
The purpose of this study is to determine if pumosetrag is effective in treating Gastroesophageal Reflux Disease (GERD) symptoms in patients who have a history of GERD symptoms and are currently taking an acid suppression therapy, such as a Proton Pump Inhibitor (PPI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with history of Gastroesophageal Reflux Disease (GERD) symptoms (heartburn, regurgitation, acid taste in mouth).
* Between ages of 18 - 70 inclusive.
* Develop GERD symptoms following ingestion of a refluxogenic meal.
* Able to take a stable Proton Pump Inhibitor (PPI) regimen for duration of study.
* Understand and sign the informed consent form.

Exclusion Criteria:

* Pregnant or lactating women.
* Allergic to pumosetrag or formulation excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Study Completion 2011-05

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Lynn Health Science Institute, Oklahoma City, Oklahoma